CLINICAL TRIAL: NCT04704011
Title: Evaluating the Impact of Basic Needs Assessment and Support to Improve Colposcopy Show Rates: The BASICS Trial
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Trial was not funded.
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 202010144
Record Dates: First submitted 2021-01-07; First posted 2021-01-11 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Colposcopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Basic Needs Assessment (Experimental): -Patients will receive a phone call from a research team member 2-4 weeks before their colposcopy appointment. The team member will remind the patient of the date and time of their appointment and conduct a basic needs assessment. Those who have at least one unmet basic need or are unsure of their current needs will be referred to the 24-hr assistance hotline, 2-1-1 United Healthy Way Missouri. After the date of their appointment, patients will be contacted to ask whether they contacted 2-1-1 and used any recommended services.
  Interventions: Other: 2-1-1 United Way Healthy Missouri Hotline; Other: National Comprehensive Cancer Network (NCCN) Distress Thermometer; Other: Basic needs survey; Other: 2-1-1 survey
- Arm 2: Usual Care Cohort (Active Comparator): -Patients will receive an automated phone call two weeks before their colposcopy appointment to remind them of the date and time of their visit.
  Interventions: Other: Usual Care Reminder Call

INTERVENTIONS:
Other: 2-1-1 United Way Healthy Missouri Hotline — This federally funded, free service connects callers with appropriate community services to help address their unmet basic needs.
  Arms: Arm 1: Basic Needs Assessment
Other: National Comprehensive Cancer Network (NCCN) Distress Thermometer — Study participants will be asked to rate the amount of distress that they have experienced in the past week (scale of 0 to 10, 10=extreme distress) and indicate areas of concern including practical basic needs and family, emotional, spiritual, and physical problems. They will also be asked to rate the amount of distress (scale 0-10) that they attribute to their abnormal cervical cancer screen.
  Arms: Arm 1: Basic Needs Assessment
Other: Basic needs survey — 11-item survey with questions regarding safety, housing, food, and financial needs
  Arms: Arm 1: Basic Needs Assessment
Other: 2-1-1 survey — This brief, 5-minute survey will be performed either in person or by phone after the participants arrive to their colposcopy appointment or after 6 weeks of their scheduled visit if they are nonadherent. The research team will ask patients regarding any changes in the status of their unmet basic needs (resolved, improved, worsened, or stayed the same) and how useful they found the 2-1-1 resource.
  Arms: Arm 1: Basic Needs Assessment
Other: Usual Care Reminder Call — -Automated phone call two weeks before their colposcopy appointment
  Arms: Arm 2: Usual Care Cohort

SUMMARY:
This randomized controlled, single-site study hopes to determine the effectiveness of a tailored phone call reminder to improve low-income patients' adherence to colposcopy.

ELIGIBILITY:
Inclusion Criteria:

* Female

  -≥ 21 years of age
* English speaking
* Able to provide verbal consent

Exclusion Criteria:

* Male
* Incarcerated
* Unable to consent
* Does not have access to a working contact phone number

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-05-31 (Estimated); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Adherence to colposcopy visit | Within 6 weeks of study enrollment

SECONDARY OUTCOMES:
Number and type of unmet basic needs as measured by Unmet Basic Needs Survey | At the time of enrollment; at least 2 weeks prior to colposcopy appointment
  -Questions asking participant about food security, housing, personal safety, neighborhood safety, sufficient money for necessities, childcare, and transportation. Scored bases on participant' self-perceived likelihood that their safety, housing, food, and financial needs would be met in the next month.
General distress scores as measured by NCCN Distress Thermometer | At the time of enrollment
  -Participant is asked to circle the number from 0-10 that best describes how much distress the participant has experienced in the past week. 0=no distress and 10=extreme distress.
Causes of distress as measured by NCCN Distress Problem List | At the time of enrollment
  -39 questions asking participant to answer yes or no to problems (practical, family, emotional, spiritual/religious, and physical) that they have experienced in the past week
Distress scores related to indications for colposcopy | At the time of enrollment
  -Score 0 (no distress) to 10 (severe distress)
Patient self-reported use of 2-1-1 services as measured by 2-1-1 Survey | After or within 1 week after colposcopy visit (estimated to be 6 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay M Kuroki, M.D., MSCI, Principal Investigator — Washington University School of Medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu